CLINICAL TRIAL: NCT01165983
Title: The Effect of Aliskiren on Endothelial Function in Pre-Diabetes and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Aristidis Veves, Rongxiang Xu, MD Professor of Surgery in the Field of Regenerative Therapeutics, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2009P000233
Record Dates: First submitted 2009-12-15; First posted 2010-07-20 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Aliskiren (Experimental)
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Placebo — 0mg tablet, taken orally for 12 weeks daily
  Arms: Placebo
Drug: Aliskiren — 150mg tablet, taken orally for 12 weeks daily
  Other Names: Trade name: Tekturna
  Arms: Aliskiren

SUMMARY:
The purpose of this research is to study and determine the effects of Aliskiren on blood vessels and blood flow. The primary hypothesis is that Aliskiren will increase endothelial function by 30% or more in comparison to the placebo group.

ELIGIBILITY:
Group 1. Subjects At Risk of Developing Type 2 Diabetes

INCLUSION CRITERIA

1. Ages of 21-80 years
2. Subjects "at risk" of developing type 2 Diabetes Mellitus (First degree relatives history of type 2 Diabetes Mellitus, History of gestational Diabetes, Known impaired glucose tolerance, Impaired fasting plasma glucose 100-126 mg/dl at the time of enrollment)

EXCLUSION CRITERIA

1. Treatment with Aliskiren (Tekturna)
2. Smokers (use of tobacco products in the previous 3 months)
3. Active or Uncontrolled Cardiovascular Disease

   * Myocardial infarction, or angina within 12 months of study participation
   * Arrhythmia (uncontrolled, highly symptomatic, requiring treatment or life-threatening)
   * CHF (Class III and IV symptoms of heart failure on less than ordinary exertion or at rest)
   * Stroke or Transient Ischemic Attack (TIA) within 12 months of study participation
   * Uncontrolled Hypertension (SBP >180 mmHg or DBP >105 mmHg; 2 abnormal readings during visit)
   * History of previous hypotensive episodes
4. Liver Disease (AST, ALT, Alk Phos levels > 2x UNL)
5. Renal Disease (creatinine > 1.7 mg/dL for women and >2.0 mg/dL for men and/or estimated GFR <30 mL/min, history of dialysis, nephrotic syndrome and known renovascular hypertension) at the time of enrollment
6. Hyperkalemia (serum potassium >5.0 meq/L)
7. Severe Dyslipidemia (TG > 600 mg/dL or Cholesterol >350 mg/dL)
8. Any Other Serious Chronic Disease Requiring Active Treatment
9. Females of Childbearing Potential Not Using an Effective Form of Birth Control as Determined by co-investigators
10. Pregnancy
11. Taking Any of the Following Medications:

    * Systemic (not inhaled) Glucocorticoids
    * Antineoplastic Agents
    * Cyclosporine, Ketoconazole, Furosemide, Warfarin
    * Bronchodilators (aminophyline, inhaled beta agonists) on a regular basis
12. Patient is known to have a history of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) and/or positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result in the past
13. History of drug or alcohol abuse within the 12months prior to dosing or evidence of such abuse as indicated by laboratory assays conducted during screening or baseline evaluations

Group 2. Type 2 Diabetic Patients

INCLUSION CRITERIA

1. Ages of 21-80 years
2. Type 2 Diabetes Mellitus stable and not expected to change during the study period

EXCLUSION CRITERIA

1. Treatment with Aliskiren (Tekturna)
2. Smokers (use of tobacco products in the previous 3 months)
3. Active or Uncontrolled Cardiovascular Disease

   * Myocardial infarction, or angina within 12 months of study participation
   * Arrhythmia (uncontrolled, highly symptomatic, requiring treatment or life-threatening)
   * CHF (Class III and IV symptoms of heart failure on less than ordinary exertion or at rest)
   * Stroke or Transient Ischemic Attack (TIA) within 12 months of study participation
   * Uncontrolled Hypertension (SBP >180 mmHg or DBP >105 mmHg; 2 abnormal readings during visit)
   * History of previous hypotensive episodes
4. Liver Disease (AST, ALT, Alk Phos levels > 2x UNL)
5. Renal Disease (creatinine > 1.7 mg/dL for women and >2.0 mg/dL for men and/or estimated GFR <30 mL/min, history of dialysis, nephrotic syndrome and known renovascular hypertension) at the time of enrollment
6. Hyperkalemia (serum potassium >5.0 meq/L)
7. Severe Dyslipidemia (TG > 600 mg/dL or Cholesterol >350 mg/dL)
8. Any Other Serious Chronic Disease Requiring Active Treatment
9. Females of Childbearing Potential Not Using an Effective Form of Birth Control as Determined by co-investigators
10. Pregnancy
11. Taking Any of the Following Medications:

    * Systemic (not inhaled) Glucocorticoids
    * Antineoplastic Agents
    * Cyclosporine, Ketoconazole, Furosemide, Warfarin
    * Bronchodilators (aminophyline, inhaled beta agonists) on a regular basis
12. Patient is known to have a history of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) and/or positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result in the past
13. History of drug or alcohol abuse within the 12months prior to dosing or evidence of such abuse as indicated by laboratory assays conducted during screening or baseline evaluations
14. Severe proliferative retinopathy that renders the subject legally blinded
15. Previous diagnosis of severe gastroparesis diabeticorum due to autonomic neuropathy that has necessitated hospital admission
16. Presence of non-healing foot ulceration due to severe peripheral diabetic neuropathy
17. Documented diabetic nephropathy manifested as macro-albuminuria, (2 of 3 urine specimens collected within a 3-6 month period with urine albumin>300 ug/mg creatinine

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-11; Primary Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aristidis Veves, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Joslin Foot Center & Microcirculation Laboratory, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Dushay JR, Tecilazich F, Kafanas A, Magargee ML, Auster ME, Gnardellis C, Dinh T, Veves A. Aliskiren improves vascular smooth muscle function in the skin microcirculation of type 2 diabetic patients with normal renal function. J Renin Angiotensin Aldosterone Syst. 2015 Jun;16(2):344-52. doi: 10.1177/1470320313489060. Epub 2013 May 13. PMID 23670354

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 124 subjects signed the ICF, but after screening procedures, 24 were found ineligible so only 100 were randomized to placebo or Aliskiren.
Period: Overall Study
Arm/Group | Placebo | Aliskiren
Started | 51 | 49
Completed | 46 | 42
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Aliskiren | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11) | 54 (11) | 54 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 30 | 50
  Male | 31 | 19 | 50
Region of Enrollment [Number; unit: participants]
  United States | 51 | 49 | 100

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Vasodilation
Description: Using ultrasound, percent change in brachial artery diameter is measured in response to an increase in shear stress from a tightened blood pressure cuff, which causes endothelium-dependent dilatation.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage change over baseline
Arm/Group | Subjects at Risk of DMII | T2DM Patients
Number analyzed (Participants) | 48 | 52
percentage change over baseline | 4.8 (0.7) | 4.4 (2.6)

2. Primary Outcome: Flow Mediated Vasodilation
Description: as for outcome 1
Time Frame: 12 Weeks post-randomization
Population: Number of subjects that completed the study
Measure: Median (Inter-Quartile Range); unit: percent change over baseline
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
percent change over baseline
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | 0.3 [-0.3 to 1.8] | 0.8 [0.3 to 2.1]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | 0.4 [0.0 to 1.0] | 0.9 [0.0 to 1.4]

3. Primary Outcome: Nitroglycerin Induced Dilation
Description: Using ultrasound, images are taken pre- and post-vasodilation of the brachial artery induced with a 0.4mg tablet of NTG.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Subjects at Risk of DMII | T2DM Patients
Number analyzed (Participants) | 48 | 52
percent change | 16.5 (4.8) | 15.2 (5.0)

4. Primary Outcome: Nitroglycerine Induced Vasodilation
Description: Using ultrasound, images are taken pre- and post-vasodilation of the brachial artery induced with a 0.4mg tablet of NTG.
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
percent change
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | 0.4 [-2.4 to 3.7] | -0.8 [-1.8 to 2.5]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | -1.4 [-3.9 to 0.4] | -0.3 [-3.4 to 1.5]

5. Primary Outcome: Skin Blood Flow Before and After Iontophoresis With Acetylcholine and Sodium Nitroprusside
Description: Laser doppler imaging is used to measure microcirculatory changes pre- and post-iontophoresis of acetylcholine and sodium nitroprusside.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: percentage change over baseline
Arm/Group | Subjects at Risk of DMII | T2DM Patients
Number analyzed (Participants) | 48 | 52
percentage change over baseline
  Acetylcholine induced skin vasodilation | 45 [19 to 62] | 38 [22 to 75]
  Sodium nitroprusside skin induced vasodilation | 38 [23 to 61] | 36 [20 to 64]

6. Primary Outcome: Skin Blood Flow Before and After Iontophoresis With Acetylcholine and Sodium Nitroprusside
Description: Laser doppler imaging is used to measure microcirculatory changes pre- and post-iontophoresis of acetylcholine (Ach) and sodium nitroprusside (NaNP).
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: percent change over baseline
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
percent change over baseline
  At risk of T2DM, Ach, Placebo n=21, Aliskiren n=20 | 6 [-31 to 37] | -1 [-43 to 15]
  At risk of T2DM, NaNP, Placebo n=21 Aliskiren n=20 | -1 [-23 to 30] | 13 [-34 to 40]
  Diabetic Patient, Ach, Placebo n=25 Aliskiren n=22 | -5 [-34 to 11] | 3 [-48 to 20]
  Diabetic Patient, NaNP, Placebo n=25 Ali. n=22 | -9 [-21 to 5] | 8 [-5 to 31]

7. Secondary Outcome: Absolute Change in Biochemical Markers of Endothelial Function, sICAM-1, ng/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
ng/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | 21 [-8 to 59] | 30 [-7 to 44]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | 13 [-25 to 45] | 14 [-13 to 40]

8. Secondary Outcome: Absolute Change in Biochemical Markers of Endothelial Function, sVCAM-1, ng/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
ng/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | 335 [-263 to 629] | 236 [-216 to 636]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | 185 [-91 to 651] | 106 [-124 to 498]

9. Secondary Outcome: Absolute Change in Biochemical Markers of Endothelial Function, t-PAI, pg/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
pg/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | 45 [-29 to 66] | 30 [-15 to 73]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | 54 [-59 to 93] | 26 [-42 to 76]

10. Secondary Outcome: Absolute Change in Biochemical Markers of Endothelial Function, C-reactive Protein, μg/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: μg/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
μg/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | -1.0 [-2.6 to 10.9] | -0.6 [-15.0 to 4.8]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | -1.7 [-17.5 to 5.5] | -2.0 [-6.0 to 0.8]

11. Secondary Outcome: Absolute Change in Biochemical Markers of Endothelial Function, E-Selectin, ng/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
ng/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | 1.9 [-1.7 to 7.1] | 0.7 [-2.1 to 11.0]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | 0.6 [-18.5 to 4.9] | -0.7 [-48.1 to 4.9]

12. Secondary Outcome: Absolute Change in Inflammatory Cytokines and Growth Factors, Osteoprotegerin, pg/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
pg/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | -36 [-78 to 80] | 97 [15 to 158]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | -24 [-86 to 75] | 48 [-24 to 127]

13. Secondary Outcome: Absolute Change in Inflammatory Cytokines and Growth Factors, Osteopontin, ng/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
ng/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | -0.3 [-5.9 to 2.1] | 2.2 [-0.8 to 4.5]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | 1.7 [-1.3 to 7.3] | 0.2 [-6.1 to 4.6]

14. Secondary Outcome: Absolute Change in Inflammatory Cytokines and Growth Factors, G-CSF, pg/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
pg/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | 1.1 [-8.5 to 13.0] | 4.0 [-0.8 to 12.8]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | 1.9 [-11.4 to 10.6] | 4.4 [-7.8 to 12.8]

15. Secondary Outcome: Absolute Change in Inflammatory Cytokines and Growth Factors, GM-CSF pg/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
pg/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | 0.4 [-1.3 to 3.7] | -0.8 [-1.4 to 4.7]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | -1.6 [-6.3 to 1.0] | 0.4 [-1.2 to 3.1]

16. Secondary Outcome: Absolute Change in Inflammatory Cytokines and Growth Factors, IL-8, pg/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
pg/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | -2.2 [-5.8 to 0.8] | -2.0 [-5.0 to 0.2]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | -2.4 [-5.9 to 1.6] | 0.6 [-2.6 to 4.0]

17. Secondary Outcome: Absolute Change in Inflammatory Cytokines and Growth Factors, MCP-1 pg/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
pg/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | -11 [-125 to 23] | -7 [-112 to 75]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | 36 [-76 to 110] | 8 [-154 to 66]

18. Secondary Outcome: Absolute Change in Inflammatory Cytokines and Growth Factors, MDC ng/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
ng/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | -0.09 [-0.32 to 0.11] | -0.07 [-0.32 to 0.08]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | -0.07 [-0.46 to 0.19] | 0.04 [-0.36 to 0.16]

19. Secondary Outcome: Absolute Change in Inflammatory Cytokines and Growth Factors, sCD-40L ng/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
ng/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | -0.8 [-3.8 to 2.7] | -3.2 [-9.6 to 4.1]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | 3.3 [-1.5 to 12.8] | -3.6 [-7.9 to 1.8]

20. Secondary Outcome: Absolute Change in Inflammatory Cytokines and Growth Factors, TNFα, pg/mL
Time Frame: 12 Weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Placebo | Aliskiren
Number analyzed (Participants) | 46 | 42
pg/mL
  At risk of T2DM, Placebo n=21, Aliskiren n=20 | -0.15 [-0.78 to 1.80] | -0.21 [-1.65 to 2.3]
  Diabetic Patients, Placebo n=25, Aliskiren n=22 | 0.30 [-3.26 to 1.67] | -0.09 [-3.20 to 1.13]

ADVERSE EVENTS:
Description: Number for "at risk" of Diabetic Ketoacidosis reduced to reflect number of subjects enrolled who were diagnosed with T2DM. Diabetic ketoacidosis is primarily a concern in patients with T1DM, however the patient who experienced ketoacidosis was later shown to have undiagnosed T1DM, improperly diagnosed as T2DM.
Arm/Group | Placebo | Aliskiren
Serious Adverse Events (participants affected / at risk) | 0/46 | 4/42
Other Adverse Events (participants affected / at risk) | 6/46 | 7/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=46) | Aliskiren (N=42)
Cardiac event (Cardiac disorders) | 0 | 2
Diabetic Ketoacidosis (Endocrine disorders) | 0/27 | 1/21
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | Aliskiren (N=42)
Constipation (Gastrointestinal disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Mild increase in Serum Calcium Level (General disorders) | 2 | 1
Decrease in Blood Glucose (Endocrine disorders) | 1 | 0
Increase in serum creatinine levels (General disorders) | 0 | 1
Numbness and cramping (Musculoskeletal and connective tissue disorders) | 1 | 1
GI virus (Gastrointestinal disorders) | 1 | 0
Decreased hematocrit (Blood and lymphatic system disorders) | 1 | 0
Bloating and gas (Gastrointestinal disorders) | 0 | 1
Increased urination (Renal and urinary disorders) | 0 | 1
Increase in eosinophil levels (Blood and lymphatic system disorders) | 0 | 1
Decrease in serum calcium (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less